CLINICAL TRIAL: NCT00282568
Title: A Phase 2, Open-Label, Multi-center Study to Assess the Pharmacokinetics, Safety and Tolerability of Tacrolimus in Stable Kidney Transplant Patients Converted From a Prograf® Based Immunosuppression Regimen to a Modified Release (MR) Tacrolimus Based Immunosuppression Regimen
Brief Title: A Study to Assess the Pharmacokinetics of a Modified-release Tacrolimus Based Immunosuppression Regimen in Stable Kidney Transplant Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 02-0-131
Record Dates: First submitted 2006-01-25; First posted 2006-01-27 (Estimated); Results first posted 2013-09-26 (Estimated); Last update posted 2013-09-26 (Estimated); Status verified 2013-07

CONDITIONS: Kidney Transplantation
Keywords: Pharmacokinetics; Therapy; Immunosuppression; Drugs, Investigational; Adult
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus Modified Release (Experimental): Participants were enrolled into the study on their stable twice-daily (bid) dose of tacrolimus on Day 1 and continued to receive a stable bid dose of tacrolimus through Day 7. Participants then converted to Tacrolimus Modified Release (MR), administered once daily at an equivalent dose to the patient's previous stable total daily dose of tacrolimus. Participants who completed the 4-week pharmacokinetic treatment period with tacrolimus MR could continue receiving tacrolimus MR as part of the extended treatment period of the study. Dose adjustments were allowed in order to maintain tacrolimus trough concentrations within the target range of 5 to 15 ng/mL and for clinical reasons.
  Interventions: Drug: Tacrolimus Modified Release (MR); Drug: tacrolimus

INTERVENTIONS:
Drug: Tacrolimus Modified Release (MR) — Oral
  Other Names: Advagraf; Astagraf XL; FK506E; FKMR; MR4
Drug: tacrolimus — Oral
  Other Names: Prograf®; FK506

SUMMARY:
A study to assess the pharmacokinetics, safety and effectiveness of tacrolimus in stable kidney transplant patients converted from a Prograf® based immunosuppression regimen to a modified release tacrolimus based immunosuppression regimen.

DETAILED DESCRIPTION:
This is a Phase II open-label, multi-center conversion study in stable, adult kidney transplant recipients to assess the pharmacokinetics, safety and effectiveness of tacrolimus in stable kidney transplant patients converted from a Prograf® based immunosuppression regimen to a modified release tacrolimus based immunosuppression regimen.

ELIGIBILITY:
Inclusion Criteria:

* Patient is currently receiving Prograf ® based immunosuppressive therapy for kidney transplantation.
* Patient has stable whole blood trough level concentrations of Prograf® and is clinically stable

Exclusion Criteria:

* Patient has previously received an organ transplant other than a kidney
* Patient is currently receiving sirolimus immunosuppression therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2002-08; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Central Contact, Study Director — Astellas Pharma US, Inc.
Locations (9):
- United States (7):
  - San Diego, California
  - Miami, Florida
  - Minneapolis, Minnesota
  - Cincinnati, Ohio
  - Portland, Oregon
  - Madison, Wisconsin
  - Milwaukee, Wisconsin
- Canada (2):
  - Edmonton, Alberta
  - Toronto, Ontario

REFERENCES:
- [Background] Alloway R, Steinberg S, Khalil K, Gourishankar S, Miller J, Norman D, Hariharan S, Pirsch J, Matas A, Zaltzman J, Wisemandle K, Fitzsimmons W, First MR. Two years postconversion from a prograf-based regimen to a once-daily tacrolimus extended-release formulation in stable kidney transplant recipients. Transplantation. 2007 Jun 27;83(12):1648-51. doi: 10.1097/01.tp.0000264056.20105.b4. PMID 17589351
- [Background] Alloway R, Steinberg S, Khalil K, Gourishankar S, Miller J, Norman D, Hariharan S, Pirsch J, Matas A, Zaltzman J, Wisemandle K, Fitzsimmons W, First MR. Conversion of stable kidney transplant recipients from a twice daily Prograf-based regimen to a once daily modified release tacrolimus-based regimen. Transplant Proc. 2005 Mar;37(2):867-70. doi: 10.1016/j.transproceed.2004.12.222. PMID 15848559

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Stable, adult kidney transplant recipients being treated with tacrolimus (Prograf)-based immunosuppressive regimen.
Pre-assignment Details: Pharmacokinetic (PK) treatment period was from Day 1 - 35. Participants who completed the PK period were eligible to continue receiving tacrolimus MR in the extended treatment period, from Day 36 up to 60 months.
Period: Pharmacokinetic Treatment Period
Arm/Group | Tacrolimus Modified Release
Started | 70
Received Tacrolimus | 68
Received Tacrolimus MR | 67
Completed | 67
Not Completed | 3
Not completed — Discontinued prior to Day 1 | 2
Not completed — Enrolled erroneously | 1
Period: Extended Treatment Period
Arm/Group | Tacrolimus Modified Release
Started | 66 (One patient who completed the PK period did not enter the extended treatment period.)
Completed | 42
Not Completed | 24
Not completed — Adverse Event | 17
Not completed — Non-compliance | 4
Not completed — Physician Decision | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Pharmacokinetic evaluable set defined as all patients with all five complete pharmacokinetic profiles (two tacrolimus and three tacrolimus MR).
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
Age Continuous [Mean (Standard Deviation); unit: years] | 46.9 (12.37)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 42
Race/Ethnicity, Customized [Number; unit: participants]
  White | 53
  Black | 12
  Asian | 1
Reason for End Stage Renal Disease [Number; unit: participants]
  Glomerulonephritis | 16
  Polycystic Kidney Disease | 8
  Hypertensive Nephrosclerosis | 6
  Immunoglobulin A Nephropathy | 6
  Diabetes | 6
  Systemic Lupus Erythematosis | 5
  Focal Segmental Glomerulonephritis | 5
  Tubular and Interstitial Disease | 3
  Unknown | 1
  Other | 10
Type of Current Transplant [Number; unit: participants]
  Cadaver | 43
  Living Related Donor | 18
  Living Nonrelated Donor | 5
Re-transplant [Number; unit: participants]
  No | 61
  Yes | 5
History of Pre-Study Dialysis [Number; unit: participants]
  No | 12
  Yes | 54

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time 0 to 24 Hours (AUC0-24) for Tacrolimus
Description: The area under the concentration-time curve was calculated from whole blood tacrolimus concentrations for both tacrolimus and tacrolimus MR at steady state using the trapezoidal rule.
Time Frame: For tacrolimus, Days 1 and 7 at 0 (pre-dose), 0.5, 1, 2, 3, 6, 8, 12 (pre-dose), 13, 14, 15, 18, 20, and 24 hours. For tacrolimus MR, Days 14 and 21 pre-dose and 0.5, 1, 2, 3, 4, 6, 8, 12, 15, 18, 20, and 24 hours post-dose.
Population: The number of participants analyzed represents the Pharmacokinetic evaluable set, defined as patients with all five complete pharmacokinetic profiles (two tacrolimus and three tacrolimus MR).
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
ng*hr/mL
  Day 1: Tacrolimus | 215.1 (59.4)
  Day 7: Tacrolimus | 206.6 (58.4)
  Day 14: Tacrolimus MR | 200.7 (57.5)
  Day 21: Tacrolimus MR | 197.6 (47.5)
Statistical Analysis 1: Comparison: Tacrolimus Modified Release; The method of analysis of variance with repeated measures was used for the comparisons of AUC0-24. Exposure at steady state was used for tacrolimus (steady state was defined as days 1 and 7) and for tacrolimus MR (steady state was defined as days 14 and 21). The natural log (ln) was used to transform AUC0-24 prior to analysis and the results were transformed back to the original scale for the presentation of results; Test type: Non-Inferiority or Equivalence — If the 90% Confidence Interval for the ratio of the natural log-transformed pharmacokinetic parameters fell within an 80% to 125% range, then the exposure between the two formulations was considered to be equivalent; Ratio of means = 94.97, 90% CI 2-sided [90.72 to 99.41] — Tacrolimus/tacrolimus MR ratio of natural log transformed means expressed as a percent

2. Secondary Outcome: Percentage of Participants With Biopsy-confirmed Acute Rejection
Description: Biopsy-confirmed acute rejection (BCAR) is defined as an episode of acute allograft rejection that was confirmed by biopsy results and was Banff grade ≥ IA. Biopsies were graded by the pathologist at the clinical site according to the 1997 Banff criteria: Borderline: No intimal arteritis present but foci of mild tubulitis; Grade I: Significant interstitial infiltration and foci of moderate to severe tubulitis; Grade II: Mild to severe intimal arteritis; Grade III: Transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic infiltrate in vessel.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
percentage of participants | 10.61 [3.18 to 18.03]

3. Primary Outcome: Maximum Observed Concentration (Cmax) of Tacrolimus
Description: The maximum concentration was calculated from whole blood tacrolimus concentrations for both tacrolimus and tacrolimus MR at steady state, without interpolation.
Time Frame: as for outcome 1
Population: The number of participants analyzed represents the Pharmacokinetic evaluable set.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
ng/mL
  Day 1: Tacrolimus | 17.2 (7.2)
  Day 7: Tacrolimus | 16.0 (6.5)
  Day 14: Tacrolimus MR | 14.3 (4.7)
  Day 21: Tacrolimus MR | 14.2 (5.1)
Statistical Analysis 1: Comparison: Tacrolimus Modified Release; The method of analysis of variance with repeated measures was used for the comparisons of Cmax. Exposure at steady state was used for tacrolimus (steady state was defined as days 1 and 7) and for tacrolimus MR (steady state was defined as days 14 and 21). The natural log (ln) was used to transform Cmax prior to analysis and the results were transformed back to the original scale for the presentation of results; Test type: Non-Inferiority or Equivalence — If the 90% CI for the ratio of the natural log-transformed pharmacokinetic parameters fell within an 80% to 125% range, then the exposure between the two formulations was considered to be equivalent; Ratio of means = 88.15, 90% CI 2-sided [82.69 to 93.96] — Tacrolimus/tacrolimus MR ratio of natural log transformed means expressed as a percent

4. Primary Outcome: Minimum Concentration of Tacrolimus (Cmin)
Description: The trough (minimum) concentration of tacrolimus determined from the tacrolimus whole blood concentration value at the 24-hour time point post- dose, prior to receiving the next dose.
Time Frame: Days 1 and 7 (tacrolimus) and Days 14 and 21 (tacrolimus MR), 24 hours post-dose.
Population: The number of participants analyzed represents the trough evaluable set defined as all patients with replicate trough measurements for both tacrolimus and tacrolimus MR.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
ng/mL
  Day 1: Tacrolimus | 6.96 (1.90)
  Day 7: Tacrolimus | 6.73 (1.99)
  Day 14: Tacrolimus MR | 6.08 (1.80)
  Day 21: Tacrolimus MR | 5.83 (1.63)
Statistical Analysis 1: Comparison: Tacrolimus Modified Release; The method of analysis of variance with repeated measures was used for the comparisons of Cmin. Exposure at steady state was used for tacrolimus (steady state was defined as days 1 and 7) and for tacrolimus MR (steady state was defined as days 14 and 21). The natural log (ln) was used to transform Cmin prior to analysis and the results were transformed back to the original scale for the presentation of results; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 3, analysis 1]; Ratio of means = 87.20, 90% CI 2-sided [82.72 to 91.93] — Tacrolimus/tacrolimus MR ratio of natural log transformed means expressed as a percent

5. Primary Outcome: Time to Maximum Observed Concentration of Tacrolimus (Tmax)
Description: The time to reach the maximum concentration of tacrolimus was calculated from whole blood tacrolimus concentrations for both tacrolimus and tacrolimus MR at steady state, without interpolation.
Time Frame: as for outcome 1
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
hours
  Day 1: Tacrolimus | 1.9 (1.8)
  Day 7: Tacrolimus | 2.0 (1.7)
  Day 14: Tacrolimus MR | 3.1 (2.3)
  Day 21: Tacrolimus MR | 2.7 (2.1)

6. Primary Outcome: Patient Survival
Description: Patient Survival defined as any participant who did not die by the time of analysis.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set, defined as all patients who took at least one dose of tacrolimus MR during the extension portion of the study.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
percentage of participants | 95.45 [90.43 to 100.00]

7. Primary Outcome: Graft Survival
Description: Graft survival was defined as any participant who did not meet the definition of graft loss, where graft loss was defined as graft failure (re-transplant or permanent return to dialysis (for more than 30 days)) or participants death.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
percentage of participants | 86.36 [78.08 to 94.64]

8. Secondary Outcome: Change From Baseline in Serum Creatinine
Description: Renal function was assessed using serum creatinine levels over the course of the study.
Time Frame: Baseline (the last day of tacrolimus on Day 7), Day 35 (end of the pharmacokinetic phase) and end of treatment (EOT; the last observed value during treatment, maximum time on study was 60 months).
Population: Modified safety analysis set defined as all patients who took at least 1 dose of tacrolimus and at least one dose of tacrolimus MR during the pharmacokinetic portion of the study. "N" indicates the number of participants with available data at each time point."
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 67
mg/dL
  Baseline [N= 67] | 1.37 (0.501)
  Change from Baseline at Day 35 [N=66] | 0.09 (0.350)
  Change from Baseline at EOT [N=67] | 0.57 (2.322)

9. Secondary Outcome: Change From Baseline in Creatinine Clearance
Description: Renal function was assessed using creatinine clearance levels calculated using the Cockcroft-Gault formula, over the course of the study.
Time Frame: as for outcome 8
Population: Modified safety analysis set
Measure: Mean (Standard Deviation); unit: mL/minute
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 67
mL/minute
  Baseline [N= 67] | 62.29 (17.531)
  Change from Baseline at Day 35 [N=66] | -2.32 (5.500)
  Change from Baseline at EOT [N=67] | -5.41 (13.335)

10. Secondary Outcome: Time to Event for Patient Non Survival
Description: For participants who died on study, the median number of days from enrollment to death due to any cause.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set who died on study.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 3
days | 1754.00 [1063.0 to 1799.0]

11. Secondary Outcome: Time to Event for Graft Non Survival
Description: For participants with graft loss, the median number of days from enrollment to graft loss. Graft loss was defined as graft failure (re-transplant or permanent return to dialysis (for more than 30 days)) or participant death.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set with graft loss.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 9
days | 1526.00 [130.0 to 2113.0]

12. Secondary Outcome: Time to First Biopsy-confirmed Acute Rejection
Description: For participants with a biopsy-confirmed acute rejection, the median number of days from enrollment to the date of biopsy confirmation. Biopsy-confirmed acute rejection (BCAR) is defined as an episode of acute allograft rejection that was confirmed by biopsy results and was Banff grade ≥ IA. Biopsies were graded by the pathologist at the clinical site according to the 1997 Banff criteria: Borderline: No intimal arteritis present but foci of mild tubulitis; Grade I: Significant interstitial infiltration and foci of moderate to severe tubulitis; Grade II: Mild to severe intimal arteritis; Grade III: Transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic infiltrate in vessel.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set with a biopsy-confirmed acute rejection.
Measure: Median (Full Range); unit: days
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 7
days | 727.00 [163.0 to 1762.0]

13. Secondary Outcome: Grade of Biopsy-confirmed Acute Rejection Episodes
Description: Biopsy-confirmed acute rejection (BCAR) is defined as an episode of acute allograft rejection that was confirmed by biopsy results and was Banff grade ≥ IA. Biopsies were graded by the pathologist at the clinical site according to the 1997 Banff criteria: Borderline: No intimal arteritis present but foci of mild tubulitis; Grade I: Significant interstitial infiltration and foci of moderate to severe tubulitis; Grade II: Mild to severe intimal arteritis; Grade III: Transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic infiltrate in vessel.
  For participants with more than one biopsy-confirmed acute rejection episode, the worst case grade is reported.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set with a biopsy-confirmed acute rejection.
Measure: Number; unit: participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 7
participants
  Grade IA | 3
  Grade IB | 1
  Grade IIA | 2
  Grade IIB | 1
  Grade III | 0

14. Secondary Outcome: Number of Participants Receiving Anti-lymphocyte Antibody Therapy for Acute Rejection
Description: Steroid-resistant rejection episodes were treated with anti-lymphocyte antibodies. If a participant had a histologically proven Banff Grade II or III rejection, they could be initiated on anti-lymphocyte antibody treatment per institutional practice. Biopsies were graded by the pathologist at the clinical site according to the 1997 Banff criteria: Borderline: No intimal arteritis present but foci of mild tubulitis; Grade I: Significant interstitial infiltration and foci of moderate to severe tubulitis; Grade II: Mild to severe intimal arteritis; Grade III: Transmural arteritis and/or arterial fibrinoid change and necrosis of medial smooth muscle cells with accompanying lymphocytic infiltrate in vessel.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
participants | 4

15. Secondary Outcome: Number of Participants With Multiple Rejection Episodes
Description: This analysis includes rejection episodes that were either confirmed by biopsy by the clinical site pathologist or were clinically treated.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
participants | 2

16. Secondary Outcome: Number of Participants With Clinically Treated Acute Rejection Episodes
Description: A clinically treated acute rejection episode was any biopsy-confirmed or suspected rejection episode that was treated with immunosuppressive therapy.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
participants | 7

17. Secondary Outcome: Number of Participants With Chronic Rejection
Description: Due to the low number of participants with biopsy-confirmed acute rejection episodes, chronic rejection was not analyzed.
Time Frame: From enrollment until the end of study (up to 60 months).
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 0

18. Secondary Outcome: Number of Participants With Treatment Failure
Description: Treatment failure was defined as discontinuation of study drug for any reason. Due to discontinuation of the study by the sponsor, treatment failure was not analyzed.
Time Frame: From enrollment until the end of study (up to 60 months).
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 0

19. Secondary Outcome: Primary Reason for Graft Loss
Description: The primary reason for graft loss was recorded by the Investigator. Graft loss was defined as graft failure (re-transplant or permanent return to dialysis) or death. GBM = glomerular basement membrane.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Participants in the modified full analysis set with graft loss.
Measure: Number; unit: participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 9
participants
  Donor GBM disease | 1
  Drug induced nephropathy | 1
  Polyoma virus | 1
  Renal insufficiency | 1
  Non-compliance with study medication | 1
  Recurrent disease | 1
  Death | 3

20. Secondary Outcome: Number of Participants Returning to Permanent Dialysis
Description: Permanent dialysis defined as dialysis for longer than 30 days.
Time Frame: From enrollment until the end of study (up to 60 months).
Population: Modified full analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 66
participants | 3

21. Secondary Outcome: Safety as Assessed by Adverse Events, Laboratory Parameters and Vital Signs
Description: An adverse event was defined as any reaction, side effect or other untoward medical occurrence, regardless of the relationship to study drug which occurred during the conduct of a clinical study. Clinically significant adverse changes in clinical status, routine laboratory studies or physical examinations were considered adverse events.
  A serious adverse event was any adverse event occurring at any dose that resulted in any of the following outcomes:
  * Death
  * Life-threatening adverse event
  * Inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability or incapacity
  * Congenital abnormality or birth defect
  * Important medical event.
Time Frame: From the first dose of tacrolimus MR formulation through the day of last dose plus 10 days (approximately 60 months).
Population: Modified safety analysis set
Measure: Number; unit: participants
Arm/Group | Tacrolimus Modified Release
Number analyzed (Participants) | 67
participants
  Any adverse event | 66
  Any serious adverse event | 39
  Adverse event leading to discontinuation | 16
  Adverse Event leading to dose changes | 29
  Death | 3

ADVERSE EVENTS:
Time Frame: From the first dose of tacrolimus MR formulation through the day of last dose plus 10 days (approximately 60 months).
Description: Adverse events are reported for the modified safety analysis set defined as all patients who took at least 1 dose of tacrolimus MR during the pharmacokinetic period of the study.
Arm/Group | Tacrolimus Modified Release
Serious Adverse Events (participants affected / at risk) | 39/67
Other Adverse Events (participants affected / at risk) | 48/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Modified Release (N=67)
Cellulitis (Infections and infestations) | 4
Escherichia urinary tract infection (Infections and infestations) | 4
Pyelonephritis (Infections and infestations) | 3
Abscess limb (Infections and infestations) | 2
Bronchitis (Infections and infestations) | 2
Urosepsis (Infections and infestations) | 2
Viral infection (Infections and infestations) | 2
Cellulitis staphylococcal (Infections and infestations) | 1
Clostridium colitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Hepatitis c (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Human polyomavirus infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Orchitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Pneumonitis cryptococcal (Infections and infestations) | 1
Pyelonephritis acute (Infections and infestations) | 1
Sepsis syndrome (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Urinary tract infection bacterial (Infections and infestations) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 2
Abdominal pain lower (Gastrointestinal disorders) | 1
Abdominal strangulated hernia (Gastrointestinal disorders) | 1
Anal ulcer (Gastrointestinal disorders) | 1
Coeliac disease (Gastrointestinal disorders) | 1
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Intestinal perforation (Gastrointestinal disorders) | 1
Palatal dysplasia (Gastrointestinal disorders) | 1
Small intestinal obstruction (Gastrointestinal disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung Nodule (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tonsil cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Renal failure acute (Renal and urinary disorders) | 7
Haematuria (Renal and urinary disorders) | 2
Renal insufficiency (Renal and urinary disorders) | 2
Glomerulonephritis focal (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Tubulointestitial nephritis (Renal and urinary disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 5
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 2
Fluid overload (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 1
Hypovolaemia (Metabolism and nutrition disorders) | 1
Arteriovenous graft site complications (Injury, poisoning and procedural complications) | 1
Complications of transplant surgery (Injury, poisoning and procedural complications) | 1
Drug toxicity (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Injury (Injury, poisoning and procedural complications) | 1
Intentional misuse (Injury, poisoning and procedural complications) | 1
Medication error (Injury, poisoning and procedural complications) | 1
Post procedural diarrhoea (Injury, poisoning and procedural complications) | 1
Renal injury (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Localised osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Aseptic necrosis bone (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1
Myopathy (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1
Chest pain (General disorders) | 2
Pyrexia (General disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 1
Malaise (General disorders) | 1
Pelvic mass (General disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Malignant hypertension (Vascular disorders) | 2
Gangrene (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Peripheral ischaemia (Vascular disorders) | 1
Angina pectoris (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Atrial Fibrillation (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Blood creatinine increased (Investigations) | 2
Weight decreased (Investigations) | 2
Anaemia (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 1
Amyloidosis (Immune system disorders) | 1
Kidney transplant rejection (Immune system disorders) | 1
Ectopic pregnancy (Pregnancy, puerperium and perinatal conditions) | 1
Vulvar Dysplasia (Reproductive system and breast disorders) | 1
Pregnancy of partner (Social circumstances) | 1
Renal transplant (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tacrolimus Modified Release (N=67)
Upper respiratory tract infection (Infections and infestations) | 18
Sinusitis (Infections and infestations) | 9
Escherichia urinary tract infection (Infections and infestations) | 8
Nasopharyngitis (Infections and infestations) | 8
Influenza (Infections and infestations) | 7
Urinary tract infection bacterial (Infections and infestations) | 6
Urinary tract infection (Infections and infestations) | 5
Herpes zoster (Infections and infestations) | 4
Pneumonia (Infections and infestations) | 4
Urinary tract infection enterococcal (Infections and infestations) | 4
Diarrhoea (Gastrointestinal disorders) | 12
Nausea (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 4
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Hypertension (Vascular disorders) | 7
Oedema Peripheral (General disorders) | 6
Blood creatinine increased (Investigations) | 6
Headache (Nervous system disorders) | 5

LIMITATIONS AND CAVEATS:
Company makes no warranties or representations of any kind as to the posting, expressed or implied, including warranties of merchantability and fitness for a particular purpose, and shall not be liable for any damages.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data or until 18 months have elapsed following study completion. Sponsor must receive a site's manuscript at least 30 days prior to publication to ensure that no confidential information of Sponsor is included in the document.